CLINICAL TRIAL: NCT00795821
Title: A Randomized, Double-Blind Comparison of LY2216684 and Placebo and Long Term Treatment With LY2216684 in Adult Patients With Major Depressive Disorder
Brief Title: A Study in Adult Patients With Major Depressive Disorder
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 11313; H9P-MC-LNBI (Other: Eli Lilly and Company)
Record Dates: First submitted 2008-11-19; First posted 2008-11-21 (Estimated); Results first posted 2018-03-20 (Actual); Last update posted 2018-03-20 (Actual); Status verified 2018-03

CONDITIONS: Depressive Disorder, Major
MeSH Terms: conditions — Depressive Disorder, Major | interventions — alpha-((5-fluoro-2-methoxyphenyl)methyl)-alpha-(tetrahydro-2H-pyran-4-yl)-2-morpholinemethanol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LY2216684 (Experimental): 10-week Acute Treatment Phase: Day after Week 0=start of 6 milligram (mg) once daily (QD) dosing; Week 1=all participants titrated to 9 mg QD; After Week 1=dose increased, maintained, or decreased to a minimum of 6 mg QD and maximum of 18 mg QD, depending on participant's tolerance of study drug.
  1-year Long-term Extension Phase: Day after Week 10=start of same LY2216684 dose participant was taking at the end of acute treatment phase; After Week 11=dose increased, maintained, or decreased to minimum of 6 mg QD and maximum of 18 mg QD based on investigator's judgment of safety and tolerability (up to Week 62).
  Interventions: Drug: LY2216684
- Placebo (Placebo Comparator): 10-week Acute Treatment Phase: 3 tablets QD for 10 weeks
  1-year Long-term Extension Phase: Day after Week 10=6 mg LY2216684 dose; After 1 week=dose escalated to 9 mg QD; After Week 11=dose increased, maintained, or decreased to minimum of 6 mg QD and maximum of 18 mg QD based on investigator's judgment of safety and tolerability (up to Week 62).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY2216684 — Flexible Dosing: 6 mg, 9 mg, 12 mg and 18 mg (3 tablets) administered QD for up to 62 weeks
  Arms: LY2216684
Drug: Placebo — Dose: 3 tablets QD for 10 weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess whether LY2216684 is superior to placebo in the treatment of adult patients with major depressive disorder.

ELIGIBILITY:
Inclusion Criteria:

* Adults age 18-65 years
* Meet criteria for major depressive disorder (MDD) as defined by Diagnostic and Statistical Manual of Mental Disorders-fourth edition-text revision (DSM-IV-TR) criteria without psychotic features
* Women of child-bearing potential must test negative for pregnancy and agree to use a reliable method of birth control
* Grid 17-item Hamilton Rating Scale for Depression (GRID-HAMD17) total score ≥18 at Visit 1 and Visit 2
* Clinical global impressions of severity (CGI-S) score ≥4 at Visit 1 and Visit 2

Exclusion Criteria:

* Are currently involved in or discontinued within the last 30 days from a clinical trial involving an off-label use of an investigational drug
* Have previously completed or withdrawn from this study or any other study investigating LY2216684
* Have had or currently have any additional ongoing DSM-IV-TR Axis 1 condition other than MDD
* Have had any anxiety disorder preceding the onset of depression that was considered the primary diagnosis within 1 year of Visit 1
* Have an Axis II disorder that would interfere with protocol compliance
* Have a current or previous diagnosis of Bipolar I or II, psychotic depression, schizophrenia, or other psychotic disorder
* Have a history of substance abuse within the past 1 year
* Women who are pregnant or breast-feeding
* Have had a lack of response of the current depressive episode to 2 or more adequate courses of antidepressant therapy, or in the judgment of the investigator, considered to have treatment-resistant depression
* Participants who are judged to be at serious suicidal risk
* Have a serious or unstable medical illness
* Have any diagnosed medical condition which could be exacerbated by noradrenergic agents including unstable hypertension, unstable heart disease, tachycardia or tachyarrhythmia, narrow angle glaucoma, or urinary hesitation or retention
* Have received treatment with a monoamine oxidase inhibitor (MAOI) within 14 days prior to Visit 1
* Have a history of severe allergies to more than 1 class of medication or multiple adverse drug reactions
* Have a history of electroconvulsive therapy (ECT), transcranial magnetic stimulation (TMS) or psychosurgery within the last year
* Have a history of any seizure disorder (other than febrile seizures)
* Require psychotropic medication other than sedative/hypnotic medication for sleep
* Have a thyroid stimulating hormone (TSH) level outside the established reference range.
* Are taking or have received treatment with any excluded medication within 7 days prior to Visit 2
* Initiation or change in intensity of psychotherapy or other non-drug therapies within 6 weeks prior to enrollment
* A positive urine drug screen for any substance of abuse at Visit 1
* Have initiated or discontinued hormone therapy within the previous 3 months prior to enrollment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 495 (Actual)
Dates: Start 2008-12; Primary Completion 2010-02 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (37):
- United States (19):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Birmingham, Alabama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Little Rock, Arkansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Beverly Hills, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cerritos, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Denver, Colorado
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hamden, Connecticut
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., North Miami, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Orlando, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., West Palm Beach, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Atlanta, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Smyrna, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Overland Park, Kansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Baltimore, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Willingboro, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Albuquerque, New Mexico
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Portland, Oregon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Memphis, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Antonio, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bellevue, Washington
- Argentina (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Buenos Aires
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., La Plata
- Finland (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Helsinki
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oulu
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tampere
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Turku
- Poland (8):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bełchatów
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bialystok
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gdansk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gorlice
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Leszno
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lublin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Torun
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tuszyn
- Russia (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kazan'
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rostov-on-Don
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint Petersburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tomsk

REFERENCES:
- [Derived] Stauffer VL, Liu P, Goldberger C, Marangell LB, Nelson C, Gorwood P, Fava M. Is the Noradrenergic Symptom Cluster a Valid Construct in Adjunctive Treatment of Major Depressive Disorder? J Clin Psychiatry. 2017 Mar;78(3):317-323. doi: 10.4088/JCP.15m09972. PMID 27685842

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The Screening Phase (Week -1 through Week 0) assessed participant eligibility for not less than 3 days and not more than 30 days. At Week 0, those participants who met entry criteria were randomized in a 1:1 ratio to either LY2216684 (dose range 6 milligram [mg] to 18 mg once daily [QD]) or placebo.
Groups:
- Placebo: 10-week Acute Treatment Phase: 3 tablets QD for 10 weeks
  1-year Long-term Extension Phase: Day after Week 10=6 mg LY2216684; After 1 week=dose escalated to 9 mg QD; After Week 11=dose increased, maintained, or decreased to minimum of 6 mg QD and maximum of 18 mg QD based on investigator's judgment of safety and tolerability (up to Week 62).
Period: Acute Treatment Phase
Arm/Group | LY2216684 | Placebo
Started | 250 | 245
Completed | 194 (4 LY-treated participants in the Acute Phase chose not to enter the Long-term Extension Phase.) | 214 (7 placebo-treated participants in the Acute Phase chose not to enter the Long-term Extension Phase.)
Not Completed | 56 | 31
Not completed — Adverse Event | 23 | 4
Not completed — Death | 1 | 0
Not completed — Lack of Efficacy | 5 | 2
Not completed — Lost to Follow-up | 9 | 12
Not completed — Physician Decision | 1 | 1
Not completed — Protocol Violation | 1 | 2
Not completed — Withdrawal by Subject | 16 | 10
Period: Long-term Extension Phase
Arm/Group | LY2216684 | Placebo
Started | 190 | 207 (All placebo-treated participants received LY2216684 in the Long-term Extension Phase.)
Completed | 100 | 115
Not Completed | 90 | 92
Not completed — Adverse Event | 25 | 32
Not completed — Lack of Efficacy | 16 | 12
Not completed — Lost to Follow-up | 20 | 16
Not completed — Physician Decision | 1 | 2
Not completed — Protocol Violation | 3 | 5
Not completed — Withdrawal by Subject | 25 | 25
Period: Taper Phase
Arm/Group | LY2216684 | Placebo
Started | 240 (N=240 participants entered Taper Phases: N=4 from Acute Phase; N=236 from Extension Phase.) | 6 (N=6 participants entered only Acute Taper Phase.)
Completed | 231 (N=231 participants completed Taper Phases: N=3 from Acute Phase; N=228 from Extension Phase.) | 6 (N=6 participants completed only Acute Taper Phase; N=0 participants entered Extension Taper Phase.)
Not Completed | 9 | 0
Not completed — Adverse Event | 2 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Physician Decision | 2 | 0
Not completed — Withdrawal by Subject | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LY2216684 | Placebo | Total
Number analyzed (Participants) | 250 | 245 | 495
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.2 (11.32) | 45.5 (11.61) | 44.8 (11.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 160 | 143 | 303
  Male | 90 | 102 | 192
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 31 | 25 | 56
  Not Hispanic or Latino | 200 | 200 | 400
  Unknown or Not Reported | 19 | 20 | 39
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 3 | 3
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 45 | 44 | 89
  White | 191 | 187 | 378
  More than one race | 9 | 7 | 16
  Unknown or Not Reported | 3 | 1 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 140 | 135 | 275
  Finland | 42 | 43 | 85
  Argentina | 13 | 13 | 26
  Poland | 44 | 45 | 89
  Russia | 11 | 9 | 20

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Montgomery-Asberg Depression Rating Scale (MADRS) at Week 10
Description: The MADRS measured severity of depressive mood symptoms. The 10-item checklist rating scale was 0 to 6, for a total score range of 0 (low severity of depressive symptoms) to 60 (high severity of depressive symptoms). Least Squares (LS) Means were adjusted for treatment, investigator, visit, treatment-by-visit, baseline score, and baseline-by-visit.
Time Frame: Baseline, Week 10
Population: The analysis population included all randomized participants with a baseline and at least 1 post-baseline value.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- LY2216684: 10-week Acute Treatment Phase: Day after Week 0=start of 6 mg QD dosing; Week 1=all participants were titrated to 9 mg QD; After Week 1=dose was increased, maintained, or decreased to a minimum of 6 mg QD and maximum of 18 mg QD, depending on participant's tolerance of study drug.
- Placebo: 10-week Acute Treatment Phase: 3 tablets QD for 10 weeks
Arm/Group | LY2216684 | Placebo
Number analyzed (Participants) | 247 | 242
units on a scale | -13.30 (0.563) | -9.82 (0.544)
Statistical Analysis 1: Comparison: LY2216684 vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Model terms included treatment, investigator, visit, treatment-by-visit, baseline score, and baseline-by-visit

2. Secondary Outcome: Mean Change From Baseline (Week 10) in Montgomery-Asberg Depression Rating Scale (MADRS) at Week 62
Description: The MADRS measured severity of depressive mood symptoms. The 10-item checklist rating scale was 0 to 6, for a total score range of 0 (low severity of depressive symptoms) to 60 (high severity of depressive symptoms). Least Squares (LS) Means were adjusted for investigator, visit, baseline score, and baseline-by-visit.
Time Frame: Baseline (Week 10), Week 62
Population: The analysis population included all participants in the Long-term Extension Phase with a baseline and at least 1 post-baseline value.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- LY2216684/LY2216684: 1-year Long-term Extension Phase: Day after Week 10=start of same LY2216684 dose participant was taking at the end of Acute Treatment Phase; After Week 11=dose increased, maintained, or decreased to minimum of 6 mg QD and maximum of 18 mg QD based on investigator's judgment of safety and tolerability (up to Week 62).
- Placebo/LY2216684: 1-year Long-term Extension Phase: Day after Week 10=6 mg LY2216684; After 1 week=dose escalated to 9 mg QD; After Week 11=dose increased, maintained, or decreased to minimum of 6 mg QD and maximum of 18 mg QD based on investigator's judgment of safety and tolerability (up to Week 62).
Arm/Group | LY2216684/LY2216684 | Placebo/LY2216684
Number analyzed (Participants) | 202 | 185
units on a scale | -7.44 (0.674) | -9.43 (0.666)

3. Secondary Outcome: Mean Change From Baseline in Sheehan Disability Scale (SDS) Global Functional Impairment at Week 10
Description: The SDS was completed by the participant and used to assess the effect of the participant's symptoms on their work/social/family life. Total of these 3 items=Global Functional Impairment score; scores ranged from 0 to 30, with higher values indicating greater disruption in the participant's work/social/family life. Least Squares (LS) Means were adjusted for treatment, investigator, visit, treatment-by-visit, baseline score, and baseline-by-visit.
Time Frame: Baseline, Week 10
Population: The analysis population included all randomized participants with a baseline and at least 1 post-baseline value.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2216684 | Placebo
Number analyzed (Participants) | 241 | 237
units on a scale | -8.21 (0.499) | -5.79 (0.484)
Statistical Analysis 1: Comparison: LY2216684 vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — To control for multiple comparisons, the analysis of this secondary outcome measure was pre-specified as a gated secondary objective. As the primary hypothesis was statistically significant, this hypothesis was tested at the 0.05 significance level; Model terms included treatment, investigator, visit, treatment-by-visit, baseline score, and baseline-by-visit

4. Secondary Outcome: Mean Change From Baseline (Week 10) in Sheehan Disability Scale (SDS) Global Functional Impairment at Week 62
Description: The SDS was completed by the participant and used to assess the effect of the participant's symptoms on their work/social/family life. Total of these 3 items=Global Functional Impairment score; scores ranged from 0 to 30, with higher values indicating greater disruption in the participant's work/social/family life. Least Squares (LS) Means were adjusted for investigator, visit, baseline score, and baseline-by-visit.
Time Frame: Baseline (Week 10), Week 62
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2216684/LY2216684 | Placebo/LY2216684
Number analyzed (Participants) | 179 | 185
units on a scale | -3.06 (0.654) | -4.56 (0.591)

5. Secondary Outcome: Mean Change From Baseline in Clinical Global Impressions of Severity (CGI-Severity) Scale at Week 10
Description: CGI-S measured severity of depression at the time of assessment. Scores ranged from 1 (normal, not at all ill) to 7 (among the most extremely ill participants). Least Squares (LS) Means were adjusted for treatment, investigator, visit, treatment-by-visit, baseline score, and baseline-by-visit.
Time Frame: Baseline, Week 10
Population: The analysis population included all randomized participants with a baseline and at least 1 post-baseline value.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2216684 | Placebo
Number analyzed (Participants) | 247 | 242
units on a scale | -1.48 (0.075) | -1.08 (0.072)
Statistical Analysis 1: Comparison: LY2216684 vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Model terms included treatment, investigator, visit, treatment-by-visit, baseline score, and baseline-by-visit

6. Secondary Outcome: Mean Change From Baseline (Week 10) in Clinical Global Impressions of Severity (CGI-Severity) Scale at Week 62
Description: CGI-S measured severity of depression at the time of assessment. Scores ranged from 1 (normal, not at all ill) to 7 (among the most extremely ill participants). Least Squares (LS) Means were adjusted for investigator, baseline score, and baseline-by-visit.
Time Frame: Baseline (Week 10), Week 62
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2216684/LY2216684 | Placebo/LY2216684
Number analyzed (Participants) | 188 | 207
units on a scale | -1.03 (0.087) | -1.24 (0.085)

7. Secondary Outcome: Mean Change From Baseline in the 16-Item Quick Inventory of Depressive Symptomatology-Self Rated (QIDS-SR16) at Week 10
Description: The QIDS-SR16 was a 16-item participant-rated measure of depressive symptomatology. The total score ranged from 0 to 27, with higher scores indicative of greater severity. Least Squares (LS) Means were adjusted for treatment, investigator, visit, treatment-by-visit, baseline score, and baseline-by-visit.
Time Frame: Baseline, Week 10
Population: The analysis population included all participants with a baseline and at least 1 post-baseline value in the Per Protocol population, defined as the subset of randomized participants who had baseline and post-baseline data collected using the correct version of the QIDS-SR16 worksheet.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2216684 | Placebo
Number analyzed (Participants) | 193 | 185
units on a scale | -6.50 (0.366) | -4.93 (0.360)
Statistical Analysis 1: Comparison: LY2216684 vs Placebo; Test type: Superiority or Other; p = 0.002, Mixed Models Analysis; Model terms included treatment, investigator, visit, treatment-by-visit, baseline score, and baseline-by-visit

8. Secondary Outcome: Mean Change From Baseline (Week 10) in the 16-Item Quick Inventory of Depressive Symptomatology-Self Rated (QIDS-SR16) at Week 62
Description: The QIDS-SR16 was a 16-item participant-rated measure of depressive symptomatology. The total score ranged from 0 to 27, with higher scores indicative of greater severity. Least Squares (LS) Means were adjusted for investigator, visit, baseline score, and baseline-by-visit.
Time Frame: Baseline (Week 10), Week 62
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Placebo/LY2216684: 1-year Long-term Extension Phase: Day after Week 10=6 mg LY2216684 dose; After 1 week=dose escalated to 9 mg QD; After Week 11=dose increased, maintained, or decreased to minimum of 6 mg QD and maximum of 18 mg QD based on investigator's judgment of safety and tolerability (up to Week 62).
Arm/Group | LY2216684/LY2216684 | Placebo/LY2216684
Number analyzed (Participants) | 183 | 203
units on a scale | -2.64 (0.422) | -3.33 (0.399)

9. Secondary Outcome: Mean Change From Baseline in the Massachusetts General Hospital Cognitive and Physical Functioning Questionnaire (CPFQ) at Week 10
Description: The CPFQ was a 7-item participant-rated questionnaire pertaining to a participant's cognitive and physical well-being. It assessed motivation, wakefulness, energy, focus, recall, word-finding difficulty, and mental acuity. Each item was scored on a 6-point scale ranging from 1 (greater than normal) to 6 (totally absent); total score ranged from 7 to 42. Least Squares (LS) Means were adjusted for treatment, investigator, and baseline score.
Time Frame: Baseline, Week 10
Population: The analysis population included all randomized participants with a baseline and at least 1 post-baseline value.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2216684 | Placebo
Number analyzed (Participants) | 241 | 238
units on a scale | -6.61 (0.435) | -5.04 (0.437)
Statistical Analysis 1: Comparison: LY2216684 vs Placebo; Test type: Superiority or Other; p = 0.007, ANCOVA; Model terms included treatment, investigator, and baseline score

10. Secondary Outcome: Mean Change From Baseline (Week 10) in the Massachusetts General Hospital Cognitive and Physical Functioning Questionnaire (CPFQ) at Week 62
Description: The CPFQ was a 7-item participant-rated questionnaire pertaining to a participant's cognitive and physical well-being. It assessed motivation, wakefulness, energy, focus, recall, word-finding difficulty, and mental acuity. Each item was scored on a 6-point scale ranging from 1 (greater than normal) to 6 (totally absent); total score ranged from 7 to 42. Least Squares (LS) Means were adjusted for investigator, visit, baseline score, and baseline-by-visit.
Time Frame: Baseline (Week 10), Week 62
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2216684/LY2216684 | Placebo/LY2216684
Number analyzed (Participants) | 180 | 188
units on a scale | -2.79 (0.534) | -3.72 (0.480)

11. Secondary Outcome: Mean Change From Baseline in the EuroQol Questionnaire-5 Dimension (EQ-5D) United States (US) Index Score at Week 10
Description: EQ-5D was a generic, multidimensional, health-related, quality of life (Qol) instrument allowing participants to rate their health state in 5 domains: mobility, self-care, usual activities, pain/discomfort, and mood. A single score between 1 and 3 was generated for each domain. For each participant, the outcome rating on the 5 domains was mapped to a single index through an algorithm. The index ranged between 0 and 1, with the higher score indicating a better health state perceived by the participant. Least Squares (LS) Means were adjusted for treatment, investigator, and baseline score.
Time Frame: Baseline, Week 10
Population: The analysis population included all randomized participants with a baseline and at least 1 post-baseline value.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2216684 | Placebo
Number analyzed (Participants) | 233 | 234
units on a scale | 0.12 (0.011) | 0.09 (0.011)
Statistical Analysis 1: Comparison: LY2216684 vs Placebo; Test type: Superiority or Other; p = 0.056, ANCOVA; Model terms included treatment, investigator, and baseline score

12. Secondary Outcome: Mean Change From Baseline (Week 10) in the EuroQol Questionnaire-5 Dimension (EQ-5D) United States (US) Index Score at Week 62
Description: EQ-5D was a generic, multidimensional, health-related, quality of life (Qol) instrument allowing participants to rate their health state in 5 domains: mobility, self-care, usual activities, pain/discomfort, mood. Single score between 1 and 3 was generated for each domain. For each participant, outcome rating on the 5 domains was mapped to a single index through an algorithm. The index ranged between 0 and 1, with higher score indicating a better health state perceived by the participant. Least Squares (LS) Means were adjusted for investigator, visit, baseline score, and baseline-by-visit.
Time Frame: Baseline (Week 10), Week 62
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2216684/LY2216684 | Placebo/LY2216684
Number analyzed (Participants) | 176 | 187
units on a scale | 0.08 (0.015) | 0.06 (0.014)

13. Secondary Outcome: Mean Change From Baseline in the Fatigue Associated With Depression (FAsD) Patient Reported Outcome (PRO): Average Score at Week 10
Description: The FAsD was a participant-rated scale with 7 items that asked how often they experience different aspects of fatigue: responses from 1 (Never) to 5 (Always); 9 items that asked how often fatigue impacts various aspects of their lives: responses from 1 (Not at all) to 5 (Very much). Average Score=mean of Items 1-5, 7-12, 14, and 16. Scores ranged from 1 to 5. Least Squares (LS) Means were adjusted for treatment, investigator, visit, treatment-by-visit, baseline score, and baseline-by-visit.
Time Frame: Baseline, Week 10
Population: The analysis population included all randomized participants with a baseline and at least 1 post-baseline value.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2216684 | Placebo
Number analyzed (Participants) | 244 | 236
units on a scale | -0.99 (0.059) | -0.74 (0.057)
Statistical Analysis 1: Comparison: LY2216684 vs Placebo; Test type: Superiority or Other; p = 0.002, Mixed Models Analysis; Model terms included treatment, investigator, visit, treatment-by-visit, baseline score, and baseline-by-visit

14. Secondary Outcome: Mean Change From Baseline (Week 10) in Fatigue Associated With Depression (FAsD) Patient Reported Outcome (PRO): Average Score at Week 62
Description: The FAsD was a participant-rated scale with 7 items that asked how often they experience different aspects of fatigue: responses from 1 (Never) to 5 (Always); 9 items that asked how often fatigue impacts various aspects of their lives: responses from 1 (Not at all) to 5 (Very much). Average Score=mean of Items 1-5, 7-12, 14, and 16. Scores ranged from 1 to 5. Least Squares (LS) Means were adjusted for investigator, visit, baseline score, and baseline-by-visit.
Time Frame: Baseline (Week 10), Week 62
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2216684/LY2216684 | Placebo/LY2216684
Number analyzed (Participants) | 184 | 207
units on a scale | -0.51 (0.076) | -0.65 (0.073)

15. Secondary Outcome: Mean Change From Baseline in the Fatigue Associated With Depression (FAsD) Patient Reported Outcome (PRO): Fatigue Experience Average Score at Week 10
Description: The FAsD was a participant-rated scale with 7 items that asked how often they experience different aspects of fatigue: responses from 1 (Never) to 5 (Always); 9 items that asked how often fatigue impacts various aspects of their lives: responses from 1 (Not at all) to 5 (Very much). Fatigue Experience Average Score=mean of Items 1 to 5, and 7. Scores ranged from 1 to 5. Least Squares (LS) Means were adjusted for treatment, investigator, visit, treatment-by-visit, baseline score, and baseline-by-visit.
Time Frame: Baseline, Week 10
Population: The analysis population included all randomized participants with a baseline and at least 1 post-baseline value.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2216684 | Placebo
Number analyzed (Participants) | 247 | 238
units on a scale | -0.96 (0.060) | -0.69 (0.058)
Statistical Analysis 1: Comparison: LY2216684 vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Model terms included treatment, investigator, visit, treatment-by-visit, baseline score, and baseline-by-visit

16. Secondary Outcome: Mean Change From Baseline (Week 10) in Fatigue Associated With Depression (FAsD) Patient Reported Outcome (PRO): Fatigue Experience Average Score at Week 62
Description: The FAsD was a participant-rated scale with 7 items that asked how often they experience different aspects of fatigue: responses from 1 (Never) to 5 (Always); 9 items that asked how often fatigue impacts various aspects of their lives: responses from 1 (Not at all) to 5 (Very much). Fatigue Experience Average Score=mean of Items 1-5, and 7. Scores ranged from 1 to 5. Least Squares (LS) Means were adjusted for investigator, visit, baseline score, and baseline-by-visit.
Time Frame: Baseline (Week 10), Week 62
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2216684/LY2216684 | Placebo/LY2216684
Number analyzed (Participants) | 186 | 207
units on a scale | -0.50 (0.080) | -0.70 (0.078)

17. Secondary Outcome: Mean Change From Baseline in the Fatigue Associated With Depression (FAsD) Patient Reported Outcome (PRO): Fatigue Impact Average Score at Week 10
Description: The FAsD was a participant-rated scale with 7 items that asked how often they experience different aspects of fatigue: responses from 1 (Never) to 5 (Always); 9 items that asked how often fatigue impacts various aspects of their lives: responses from 1 (Not at all) to 5 (Very much). Fatigue Impact Average Score=mean of Items 8-12, 14, and 16. Scores ranged from 1 to 5. Least Squares (LS) Means were adjusted for treatment, investigator, visit, treatment-by-visit, baseline score, and baseline-by-visit.
Time Frame: Baseline, Week 10
Population: The analysis population included all randomized participants with a baseline and at least 1 post-baseline value.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2216684 | Placebo
Number analyzed (Participants) | 244 | 240
units on a scale | -1.02 (0.062) | -0.77 (0.060)
Statistical Analysis 1: Comparison: LY2216684 vs Placebo; Test type: Superiority or Other; p = 0.003, Mixed Models Analysis; Model terms included treatment, investigator, visit, treatment-by-visit, baseline score, and baseline-by-visit

18. Secondary Outcome: Mean Change From Baseline (Week 10) in Fatigue Associated With Depression (FAsD) Patient Reported Outcome (PRO): Fatigue Impact Average Score at Week 62
Description: The FAsD was a participant-rated scale with 7 items that asked how often they experience different aspects of fatigue: responses from 1 (Never) to 5 (Always); 9 items that asked how often fatigue impacts various aspects of their lives: responses from 1 (Not at all) to 5 (Very much). Fatigue Impact Average Score=mean of Items 8-12, 14, and 16. Scores ranged from 1 to 5. Least Squares (LS) Means were adjusted for investigator, visit, baseline score, and baseline-by-visit.
Time Frame: Baseline (Week 10), Week 62
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- LY2216684: 1-year Long-term Extension Phase: Day after Week 10=start of same LY2216684 dose participant was taking at the end of Acute Treatment Phase; After Week 11=dose increased, maintained, or decreased to minimum of 6 mg QD and maximum of 18 mg QD based on investigator's judgment of safety and tolerability (up to Week 62).
- Placebo: 1-year Long-term Extension Phase: Day after Week 10=6 mg LY2216684; After 1 week=dose escalated to 9 mg QD; After Week 11=dose increased, maintained, or decreased to minimum of 6 mg QD and maximum of 18 mg QD based on investigator's judgment of safety and tolerability (up to Week 62).
Arm/Group | LY2216684 | Placebo
Number analyzed (Participants) | 185 | 207
units on a scale | -0.51 (0.078) | -0.58 (0.081)

19. Secondary Outcome: Mean Change From Baseline in the Brief Fatigue Inventory (BFI) Global Total Score at Week 10
Description: The BFI was a participant-rated scale consisting of 9 items: 3 items assessed severity of fatigue at its "worst," "usual," and "now" during normal waking hours: 0=no fatigue to 10=fatigue as bad as you can imagine; 6 items assessed the degree to which fatigue has interfered with different aspects of the participant's life during the past 24 hours: 0=does not interfere to 10=completely interferes. The BFI Global Total Score was the mean of the 9 item scores and ranged from 0 to 10. Least Squares (LS) Means were adjusted for treatment, investigator, and baseline score.
Time Frame: Baseline, Week 10
Population: The analysis population included all randomized participants with a baseline and at least 1 post-baseline value.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2216684 | Placebo
Number analyzed (Participants) | 241 | 237
units on a scale | -2.25 (0.147) | -1.74 (0.148)
Statistical Analysis 1: Comparison: LY2216684 vs Placebo; Test type: Superiority or Other; p = 0.009, ANCOVA; Model terms included treatment, investigator, and baseline score

20. Secondary Outcome: Mean Change From Baseline (Week 10) in Brief Fatigue Inventory (BFI) Global Total Score at Week 62
Description: The BFI was a participant-rated scale consisting of 9 items: 3 items assessed severity of fatigue at its "worst," "usual," and "now" during normal waking hours: 0=no fatigue to 10=fatigue as bad as you can imagine; 6 items assessed the degree to which fatigue has interfered with different aspects of the participant's life during the past 24 hours: 0=does not interfere to 10=completely interferes. The BFI Global Total Score was the mean of the 9 item scores and ranged from 0 to 10. Least Squares (LS) Means were adjusted for investigator, visit, baseline score, and baseline-by-visit.
Time Frame: Baseline (Week 10), Week 62
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2216684/LY2216684 | Placebo/LY2216684
Number analyzed (Participants) | 180 | 188
units on a scale | -1.28 (0.202) | -1.59 (0.187)

21. Secondary Outcome: Mean Change From Baseline in the Visual Analogue Scale for Fatigue (VAS-F) Overall Severity and Interference With Daily Activities Scores at Week 10
Description: The VAS-F was a self-rated assessment with 2 items. For the Overall Severity of Fatigue item, the participant placed a vertical mark on a 100-millimeter (mm) line between 2 anchors (0=not at all to 100=as severe as I can imagine). For the Interference With Daily Activities Due to Fatigue item, the participant placed a vertical mark on a 100 mm line between 2 anchors (0=not at all to 100=complete disability [unable to do any activities]). Least Squares (LS) Means were adjusted for treatment, investigator, visit, treatment-by-visit, baseline score, and baseline-by-visit.
Time Frame: Baseline, Week 10
Population: The analysis population included all randomized participants with a baseline and at least 1 post-baseline value.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2216684 | Placebo
Number analyzed (Participants) | 247 | 242
units on a scale
  Severity of Overall Fatigue | -23.30 (1.813) | -16.69 (1.757)
  Fatigue Interference With Daily Activities | -24.48 (1.831) | -18.62 (1.775)
Statistical Analysis 1: Comparison: LY2216684 vs Placebo; Test type: Superiority or Other; p = 0.008, Mixed Models Analysis — P-value for Severity of Overall Fatigue; Model terms included treatment, investigator, visit, treatment-by-visit, baseline score, and baseline-by-visit
Statistical Analysis 2: Comparison: LY2216684 vs Placebo; Test type: Superiority or Other; p = 0.024, Mixed Models Analysis — P-value for Fatigue Interference with Daily Activities; Model terms included treatment, investigator, visit, treatment-by-visit, baseline score, and baseline-by-visit

22. Secondary Outcome: Mean Change From Baseline (Week 10) in the Visual Analogue Scale for Fatigue (VAS-F) Overall Severity and Interference With Daily Activities Scores at Week 62
Description: The VAS-F was a self-rated assessment with 2 items. For the Overall Severity of Fatigue item, the participant placed a vertical mark on a 100-millimeter (mm) line between 2 anchors (0=not at all to 100=as severe as I can imagine). For the Interference With Daily Activities Due to Fatigue item, the participant placed a vertical mark on a 100 mm line between 2 anchors (0=not at all to 100=complete disability [unable to do any activities]). Least Squares (LS) Means were adjusted for investigator, visit, baseline score, and baseline-by-visit.
Time Frame: Baseline (Week 10), Week 62
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2216684/LY2216684 | Placebo/LY2216684
Number analyzed (Participants) | 187 | 206
units on a scale
  Overall Severity of Fatigue | -12.72 (2.277) | -18.69 (1.990)
  Fatigue Interference With Daily Activities | -13.89 (2.229) | -17.47 (1.996)

23. Secondary Outcome: Percentage of Participants Reporting Resource Utilization at Week 10
Description: The Resource Utilization form assessed the frequency and type of medical services that participants have used within the last year, or since the last visit. Resources reported by at least 5% of participants in either treatment group were provided.
Time Frame: Baseline through Week 10
Population: The analysis population included all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | LY2216684 | Placebo
Number analyzed (Participants) | 226 | 229
percentage of participants
  Use of Primary Doctor | 13.3 | 10.9
  Use of Specialist | 5.8 | 5.7
  Other Diagnostic Tests | 6.6 | 5.7
  Prescribed Medication | 34.1 | 29.3
Statistical Analysis 1: Comparison: LY2216684 vs Placebo; Test type: Superiority or Other; p = 0.261, Cochran-Mantel-Haenszel — P-value for participants reporting use of primary doctor; Cochran-Mantel-Haenszel (CMH) test controlling for investigator
Statistical Analysis 2: Comparison: LY2216684 vs Placebo; Test type: Superiority or Other; p = 0.868, Cochran-Mantel-Haenszel — P-value for participants reporting use of specialist; Cochran-Mantel-Haenszel (CMH) test controlling for investigator
Statistical Analysis 3: Comparison: LY2216684 vs Placebo; Test type: Superiority or Other; p = 0.495, Cochran-Mantel-Haenszel — P-value for participants reporting other diagnostic tests; Cochran-Mantel-Haenszel (CMH) test controlling for investigator
Statistical Analysis 4: Comparison: LY2216684 vs Placebo; Test type: Superiority or Other; p = 0.189, Cochran-Mantel-Haenszel — P-value for participants reporting prescribed medication; Cochran-Mantel-Haenszel (CMH) test controlling for investigator

24. Secondary Outcome: Percentage of Participants Reporting Resource Utilization at Week 62
Description: as for outcome 23
Time Frame: Baseline (Week 10) through Week 62
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | LY2216684/LY2216684 | Placebo/LY2216684
Number analyzed (Participants) | 172 | 180
percentage of participants
  Use of Primary Doctor | 27.3 | 24.4
  Use of Specialist | 14.0 | 13.3
  Use of ER or Urgent Care: Other Reason | 5.8 | 5.6
  Special Scans/Tests | 5.2 | 3.3
  Other Diagnostic Tests | 19.2 | 15.6
  Prescribed Medications | 39.5 | 35.0

25. Secondary Outcome: Percentage of Participants With Suicidal Ideation, Behavior, and Acts Based on The Columbia Suicide Severity Rating Scale (C-SSRS) at Week 10
Description: C-SSRS scale captured occurrence, severity, and frequency of suicide-related thoughts and behaviors. Number of participants with suicidal ideation, behavior, and acts were provided. Suicidal ideation=a "yes" answer to any 1 of 5 suicidal ideation questions (including wish to be dead) and 4 different categories of active suicidal ideation. Suicidal behavior=a "yes" answer to any of 5 suicidal behavior questions: preparatory acts or behavior, aborted attempt, interrupted attempt, actual attempt, and completed suicide. Suicidal act=a "yes" answer to actual attempt or completed suicide.
Time Frame: Baseline through Week 10
Population: The analysis population included all randomized participants with a baseline and at least 1 post-baseline C-SSRS value.
Measure: Number; unit: percentage of participants
Arm/Group | LY2216684 | Placebo
Number analyzed (Participants) | 247 | 242
percentage of participants
  Suicidal ideation | 7.3 | 8.3
  Suicidal behavior | 0.0 | 0.0
  Suicidal acts | 0.0 | 0.0
Statistical Analysis 1: Comparison: LY2216684 vs Placebo; Test type: Superiority or Other; p = 0.737, Fisher Exact — P-value for suicidal ideation

26. Secondary Outcome: Percentage of Participants With Suicidal Ideation, Behavior, and Acts Based on The Columbia Suicide Severity Rating Scale (C-SSRS) at Week 62
Description: as for outcome 25
Time Frame: Baseline (Week 10) through Week 62
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | LY2216684/LY2216684 | Placebo/LY2216684
Number analyzed (Participants) | 188 | 207
percentage of participants
  Suicidal ideation | 5.9 | 6.8
  Suicidal behavior | 1.1 | 0.5
  Suicidal acts | 0.0 | 0.5

27. Secondary Outcome: Mean Change From Baseline in Supine Systolic and Diastolic Blood Pressure at Week 10
Description: Blood pressure was collected while the participant was in the supine position. Least Squares (LS) Means were adjusted for treatment, investigator, visit, treatment-by-visit, baseline score, and baseline-by-visit.
Time Frame: Baseline, Week 10
Population: The analysis population included all randomized participants with a baseline and at least 1 post-baseline value.
Measure: Least Squares Mean (Standard Error); unit: millimeters of mercury (mm Hg)
Arm/Group | LY2216684 | Placebo
Number analyzed (Participants) | 246 | 242
millimeters of mercury (mm Hg)
  Supine systolic | 1.45 (0.708) | -1.57 (0.683)
  Supine diastolic | 3.54 (0.527) | -0.64 (0.510)
Statistical Analysis 1: Comparison: LY2216684 vs Placebo; Test type: Superiority or Other; p = 0.002, Mixed Models Analysis — P-value for change in supine systolic blood pressure; Model terms included treatment, investigator, visit, treatment-by-visit, baseline score, and baseline-by-visit
Statistical Analysis 2: Comparison: LY2216684 vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — P-value for change in supine diastolic blood pressure; Model terms included treatment, investigator, visit, treatment-by-visit, baseline score, and baseline-by-visit

28. Secondary Outcome: Mean Change From Baseline (Week 10) in Supine Systolic and Diastolic Blood Pressure at Week 62
Description: Blood pressure was collected while the participant was in the supine position. Least Squares (LS) Means were adjusted for investigator, visit, baseline score, and baseline-by-visit.
Time Frame: Baseline (Week 10), Week 62
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: millimeters of mercury (mm Hg)
Arm/Group | LY2216684/LY2216684 | Placebo/LY2216684
Number analyzed (Participants) | 188 | 207
millimeters of mercury (mm Hg)
  Supine systolic | 0.52 (1.017) | 2.55 (1.064)
  Supine diastolic | -0.68 (0.724) | 2.25 (0.710)

29. Secondary Outcome: Mean Change From Baseline in Supine Pulse at Week 10
Description: Pulse was collected while the participant was in the supine position. Least Squares (LS) Means were adjusted for treatment, investigator, visit, treatment-by-visit, baseline score, and baseline-by-visit.
Time Frame: Baseline, Week 10
Population: The analysis population included all randomized participants with a baseline and at least 1 post-baseline value.
Measure: Least Squares Mean (Standard Error); unit: beats per minute (bpm)
Arm/Group | LY2216684 | Placebo
Number analyzed (Participants) | 246 | 242
beats per minute (bpm) | 9.72 (0.677) | -0.11 (0.655)
Statistical Analysis 1: Comparison: LY2216684 vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Model terms included treatment, investigator, visit, treatment-by-visit, baseline score, and baseline-by-visit

30. Secondary Outcome: Mean Change From Baseline (Week 10) in Supine Pulse at Week 62
Description: Pulse was collected while the participant was in the supine position. Least Squares (LS) Means were adjusted for investigator, visit, baseline score, and baseline-by-visit.
Time Frame: Baseline (Week 10), Week 62
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: beats per minute (bpm)
Arm/Group | LY2216684/LY2216684 | Placebo/LY2216684
Number analyzed (Participants) | 188 | 207
beats per minute (bpm) | -1.15 (0.970) | 7.33 (0.875)

31. Secondary Outcome: Pharmacokinetic (PK) Parameter: Plasma Concentration of LY2216684
Description: Blood samples collected from participants that received LY2216684 were measured to determine the plasma LY2216684 concentrations.
Time Frame: Baseline through Week 62
Population: N=number of participants analyzed (N=365); n=number of plasma LY2216684 concentration observations. The sum of the individual 'n' values for each dose group does not equal 365 since the same participant could have received various doses during his/her participation in the study.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Groups:
- LY2216684: 10-week Acute Treatment Phase: Day after Week 0=start of 6 mg QD dosing; Week 1=all participants were titrated to 9 mg QD; After Week 1=dose was increased, maintained, or decreased to a minimum of 6 mg QD and maximum of 18 mg QD, depending on participant's tolerance of study drug.
  1-year Long-term Extension Phase: Day after Week 10=start of same LY2216684 dose participant was taking at the end of acute treatment phase, or 6 mg LY2216684 dose if participants were taking placebo; After Week 1=dose escalated to 9 mg QD; After Week 11=dose increased, maintained, or decreased to minimum of 6 mg QD and maximum of 18 mg QD based on investigator's judgment of safety and tolerability (up to Week 62).
Arm/Group | LY2216684
Number analyzed (Participants) | 365
nanograms per milliliter (ng/mL)
  6 mg LY2216684: number analyzed (Participants) | 162
  6 mg LY2216684 | 12.3 (8.55)
  9 mg LY2216684: number analyzed (Participants) | 328
  9 mg LY2216684 | 18.2 (13.6)
  12 mg LY2216684: number analyzed (Participants) | 136
  12 mg LY2216684 | 26.0 (17.3)
  18 mg LY2216684: number analyzed (Participants) | 185
  18 mg LY2216684 | 40.0 (25.5)

ADVERSE EVENTS:
Groups:
- LY2216684 - Acute: 10-week Acute Treatment Phase: Day after Week 0=start of 6 milligram (mg) once daily (QD) dosing; Week 1=all participants titrated to 9 mg QD; After Week 1=dose increased, maintained, or decreased to a minimum of 6 mg QD and maximum of 18 mg QD, depending on participant's tolerance of study drug.
- Placebo - Acute: 10-week Acute Treatment Phase: 3 tablets QD for 10 weeks
- LY2216684/LY2216684 - Extension: 1-year Long-term Extension Phase: Day after Week 10=start of same LY2216684 dose participant was taking at the end of Acute Treatment Phase; After Week 11=dose increased, maintained, or decreased to minimum of 6 mg QD and maximum of 18 mg QD based on investigator's judgment of safety and tolerability (up to Week 62).
- Placebo/LY2216684 - Extension: 1-year Long-term Extension Phase: Day after Week 10=6 mg LY2216684; After 1 week=dose escalated to 9 mg QD; After Week 11=dose increased, maintained, or decreased to minimum of 6 mg QD and maximum of 18 mg QD based on investigator's judgment of safety and tolerability (up to Week 62).
- LY2216684 - Taper: Participants who took 18 mg LY2216684 received 12 mg QD for 1 week followed by 6 mg QD for 1 week. Participants who took 12 mg, 9 mg, or 6 mg LY2216684 received 6 mg QD for 2 weeks.
- Placebo - Taper: Participants who took placebo remained on placebo for 2 weeks.
Arm/Group | LY2216684 - Acute | Placebo - Acute | LY2216684/LY2216684 - Extension | Placebo/LY2216684 - Extension | LY2216684 - Taper | Placebo - Taper
Serious Adverse Events (participants affected / at risk) | 2/250 | 2/245 | 6/190 | 5/207 | 0/240 | 0/6
Other Adverse Events (participants affected / at risk) | 171/250 | 133/245 | 126/190 | 155/207 | 15/240 | 0/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | LY2216684 - Acute (N=250) | Placebo - Acute (N=245) | LY2216684/LY2216684 - Extension (N=190) | Placebo/LY2216684 - Extension (N=207) | LY2216684 - Taper (N=240) | Placebo - Taper (N=6)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tachycardia paroxysmal (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intentional overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lumbar radiculopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ruptured cerebral aneurysm (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abortion missed (Pregnancy, puerperium and perinatal conditions) | 1/160 (1) | 0/143 (0) | 0/120 (0) | 0/120 (0) | 0/143 (0) | 0/2 (0)
Drug abuse (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Major depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Schizoaffective disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | LY2216684 - Acute (N=250) | Placebo - Acute (N=245) | LY2216684/LY2216684 - Extension (N=190) | Placebo/LY2216684 - Extension (N=207) | LY2216684 - Taper (N=240) | Placebo - Taper (N=6)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Macrocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aortic valve sclerosis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrioventricular block first degree (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bundle branch block right (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac flutter (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Left atrial dilatation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 6 (7) | 2 (4) | 2 (2) | 8 (10) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 12 (13) | 2 (2) | 8 (9) | 17 (21) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Eye disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye pruritus (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye swelling (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lacrimation increased (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Photophobia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Retinal tear (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 5 (5) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (3) | 6 (7) | 0 (0) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 5 (7) | 4 (5) | 1 (1) | 5 (5) | 0 (0) | 0 (0)
Bowel movement irregularity (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 18 (18) | 6 (6) | 6 (7) | 12 (13) | 2 (2) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 10 (11) | 2 (2) | 5 (5) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 11 (13) | 9 (9) | 8 (9) | 5 (5) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 4 (5) | 5 (5) | 4 (5) | 3 (3) | 1 (1) | 0 (0)
Epigastric discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 3 (3) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (2) | 1 (2) | 0 (0) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 39 (40) | 12 (14) | 13 (15) | 23 (29) | 1 (1) | 0 (0)
Paraesthesia oral (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 3 (3) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 9 (9) | 1 (2) | 3 (3) | 6 (6) | 0 (0) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 2 (2) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Device leakage (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 7 (7) | 5 (5) | 1 (1) | 5 (5) | 1 (1) | 0 (0)
Feeling abnormal (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Feeling cold (General disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Feeling drunk (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Feeling hot (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Feeling jittery (General disorders) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Feeling of body temperature change (General disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hunger (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Irritability (General disorders) | 9 (10) | 10 (10) | 3 (3) | 2 (2) | 2 (2) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Medical device complication (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sluggishness (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thirst (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vessel puncture site haematoma (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gallbladder disorder (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Abscess limb (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 4 (4) | 3 (3) | 6 (6) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cervicitis (Infections and infestations) | 0/160 (0) | 0/143 (0) | 1/120 (1) | 0/120 (0) | 0/143 (0) | 0/2 (0)
Chlamydial infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Croup infectious (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fungal infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Groin abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infected bites (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infectious mononucleosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 1 (1) | 2 (2) | 3 (4) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Measles (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 11 (11) | 7 (7) | 7 (7) | 18 (18) | 0 (0) | 0 (0)
Oral fungal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulpitis dental (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 7 (7) | 3 (3) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Sinusitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Streptococcal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tinea pedis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tinea versicolour (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 6 (6) | 9 (9) | 10 (12) | 10 (11) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2) | 2 (2) | 4 (4) | 0 (0) | 0 (0)
Vaginal infection (Infections and infestations) | 0/160 (0) | 1/143 (1) | 1/120 (1) | 0/120 (0) | 0/143 (0) | 0/2 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Vulvovaginal mycotic infection (Infections and infestations) | 1/160 (1) | 0/143 (0) | 0/120 (0) | 0/120 (0) | 0/143 (0) | 0/2 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Arthropod sting (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Drug exposure during pregnancy (Injury, poisoning and procedural complications) | 1/160 (1) | 0/143 (0) | 0/120 (0) | 1/120 (1) | 0/143 (0) | 0/2 (0)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Joint sprain (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Scapula fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal cord injury sacral (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sunburn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bleeding time prolonged (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 3 (3) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood pressure diastolic decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood pressure diastolic increased (Investigations) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 11 (11) | 7 (8) | 7 (7) | 8 (8) | 0 (0) | 0 (0)
Blood pressure orthostatic decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Blood pressure orthostatic increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood pressure systolic increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Heart rate decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Heart rate increased (Investigations) | 16 (16) | 4 (4) | 9 (9) | 13 (14) | 1 (1) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Transaminases increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tuberculin test positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 3 (3) | 1 (1) | 4 (4) | 1 (1) | 0 (0) | 0 (0)
Weight increased (Investigations) | 4 (4) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 11 (11) | 3 (3) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Increased appetite (Metabolism and nutrition disorders) | 3 (3) | 3 (3) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3) | 5 (6) | 2 (2) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (3) | 4 (5) | 3 (3) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Joint crepitation (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 4 (4) | 1 (1) | 0 (0) | 0 (0)
Neck mass (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 3 (3) | 5 (5) | 0 (0) | 0 (0)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sensation of heaviness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tenosynovitis stenosans (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Amnesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aphasia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Complex regional pain syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Crying (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Disturbance in attention (Nervous system disorders) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 17 (18) | 3 (4) | 4 (4) | 9 (10) | 0 (0) | 0 (0)
Dizziness exertional (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness postural (Nervous system disorders) | 3 (3) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Drug withdrawal headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Head titubation (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 27 (37) | 22 (28) | 16 (21) | 27 (32) | 1 (1) | 0 (0)
Hypersomnia (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Hypogeusia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokinesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intercostal neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Memory impairment (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mental impairment (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nerve compression (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 4 (4) | 1 (1) | 4 (4) | 4 (6) | 0 (0) | 0 (0)
Parosmia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Poor quality sleep (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sedation (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Sinus headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 10 (13) | 7 (7) | 3 (4) | 7 (7) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Tension headache (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0/160 (0) | 0/143 (0) | 1/120 (1) | 0/120 (0) | 0/143 (0) | 0/2 (0)
Abnormal dreams (Psychiatric disorders) | 2 (2) | 1 (1) | 1 (1) | 5 (5) | 0 (0) | 0 (0)
Aggression (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Anorgasmia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 2 (4) | 6 (7) | 5 (5) | 3 (3) | 0 (0) | 0 (0)
Binge eating (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blunted affect (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bruxism (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depressed mood (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dissociation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Emotional disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Euphoric mood (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Initial insomnia (Psychiatric disorders) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 16 (17) | 9 (9) | 9 (9) | 14 (14) | 0 (0) | 0 (0)
Libido decreased (Psychiatric disorders) | 7 (7) | 0 (0) | 2 (2) | 3 (4) | 0 (0) | 0 (0)
Loss of libido (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Middle insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Mood swings (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nervousness (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nicotine dependence (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nightmare (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Orgasm abnormal (Psychiatric disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Orgasmic sensation decreased (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Panic attack (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Restlessness (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Sleep disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tension (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Terminal insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tobacco withdrawal symptoms (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 3 (3) | 0 (0) | 1 (1) | 7 (7) | 0 (0) | 0 (0)
Micturition urgency (Renal and urinary disorders) | 2 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Nephritis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nocturia (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal cyst (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urethral pain (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary hesitation (Renal and urinary disorders) | 6 (6) | 1 (1) | 5 (6) | 5 (5) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract disorder (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urine flow decreased (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urine odour abnormal (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Adnexa uteri pain (Reproductive system and breast disorders) | 1/160 (1) | 0/143 (0) | 0/120 (0) | 0/120 (0) | 0/143 (0) | 0/2 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 0/160 (0) | 0/143 (0) | 1/120 (1) | 0/120 (0) | 0/143 (0) | 0/2 (0)
Ejaculation disorder (Reproductive system and breast disorders) | 2/90 (2) | 0/102 (0) | 1/70 (1) | 0/87 (0) | 0/97 (0) | 0/4 (0)
Ejaculation failure (Reproductive system and breast disorders) | 0/90 (0) | 0/102 (0) | 0/70 (0) | 2/87 (2) | 0/97 (0) | 0/4 (0)
Epididymitis (Reproductive system and breast disorders) | 1/90 (1) | 0/102 (0) | 0/70 (0) | 0/87 (0) | 0/97 (0) | 0/4 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 9/90 (10) | 1/102 (1) | 1/70 (1) | 9/87 (9) | 0/97 (0) | 0/4 (0)
Nipple disorder (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oligomenorrhoea (Reproductive system and breast disorders) | 1/160 (1) | 0/143 (0) | 0/120 (0) | 0/120 (0) | 0/143 (0) | 0/2 (0)
Ovarian cyst (Reproductive system and breast disorders) | 0/160 (0) | 1/143 (1) | 0/120 (0) | 1/120 (1) | 0/143 (0) | 0/2 (0)
Penile pain (Reproductive system and breast disorders) | 1/90 (1) | 0/102 (0) | 0/70 (0) | 0/87 (0) | 0/97 (0) | 0/4 (0)
Penis disorder (Reproductive system and breast disorders) | 0/90 (0) | 0/102 (0) | 0/70 (0) | 1/87 (1) | 0/97 (0) | 0/4 (0)
Prostatomegaly (Reproductive system and breast disorders) | 0/90 (0) | 0/102 (0) | 1/70 (1) | 0/87 (0) | 0/97 (0) | 0/4 (0)
Scrotal pain (Reproductive system and breast disorders) | 1/90 (1) | 0/102 (0) | 2/70 (3) | 0/87 (0) | 0/97 (0) | 0/4 (0)
Testicular pain (Reproductive system and breast disorders) | 1/90 (1) | 0/102 (0) | 0/70 (0) | 1/87 (1) | 0/97 (0) | 0/4 (0)
Uterine haemorrhage (Reproductive system and breast disorders) | 0/160 (0) | 1/143 (1) | 0/120 (0) | 0/120 (0) | 0/143 (0) | 0/2 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 4 (5) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal blistering (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Yawning (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 14 (14) | 4 (4) | 12 (12) | 28 (37) | 1 (1) | 0 (0)
Hypoaesthesia facial (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Piloerection (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin warm (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ex-tobacco user (Social circumstances) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Angiopathy (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 5 (6) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 6 (6) | 2 (2) | 2 (2) | 5 (5) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral coldness (Vascular disorders) | 5 (5) | 2 (2) | 3 (3) | 3 (3) | 0 (0) | 0 (0)
Poor peripheral circulation (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vasoconstriction (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days